## Suppressive Antibacterial Therapy with Once-weekly Solosec® (secnidazole) Oral Granules to Prevent Recurrent Bacterial Vaginosis

Drug Name: Solosec® (secnidazole) Oral Granules, 2 g

NCT # 05033743

**Document Date: 02/17/2023** 

Chemen M. Neal MD, Associate Professor
Department of Obstetrics & Gynecology

550 N. University Ave Suite 2440

Indianapolis, IN 46202

## 1.1. Statistical Methods

To assess the efficacy of secnidazole, we estimated failure rates and 95% exact confidence intervals for initial treatment, suppression therapy following initial resolution of BV symptoms, and overall. For the time-to-failure analysis, time was defined as the number of days since the second visit where clinical resolution of initial BV was confirmed. The non-parametric maximum likelihood estimate (NPMLE) of the survival curve was estimated using the interval package in R to account for the interval censored data. Results are presented using an Amsel criteria score of  $\geq 3$  as well as  $\geq 1$  for BV diagnosis. All analyses were conducted using R 4.2.2 (R Core Team, 2020) in RStudio (RStudio Team 2021).